CLINICAL TRIAL: NCT00588445
Title: Phase II Trial to Correlate Radiographic Response Induced By Gefitinib With Mutations in the Protein-Tyrosine Kinase Domain of the EGF Receptor Gene in Patients With NSCLC
Brief Title: Phase II Trial to Correlate Radiographic Response Induced By Gefitinib With Mutations in the Protein-Tyrosine Kinase Domain of the EGF Receptor Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-071; CA113653
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer; Bronchioloalveolar Cancer
Keywords: Lung Cancer; Non-small cell lung cancer; Gefitnib; Cancer; NSCLC; bronchioloalveolar cancer; smoker
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Gefitinib

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Patients will receive gefitinib 250 mg po daily for at least 21 days preoperatively (depending on the timing of the surgery). Treatment with gefitinib will be stopped 2 days before the date of surgery.
  Patients who have had at least a minor response to gefitinib therapy preoperatively (> 25% reduction in tumor measured bidimensionally) and / or have mutations in the protein-tyrosine kinase domain of the EGF receptor gene identified will continue on the study and will resume gefitinib treatment after at least 7 days from surgery providing adequate wound healing has occurred.
  Patients who are determined to be candidates for adjuvant chemotherapy and/or radiation therapy by their treating physician may receive treatment with adjuvant chemotherapy and/or radiation therapy. The post-operative gefitinib will be started after completion of the chemotherapy and/or radiation therapy.

SUMMARY:
The purpose of this research study is to:

* see if gefitinib pills can shrink Stage 1 or 2 non-small cell lung cancers before surgery
* see if your non-small cell lung cancer has a mutation in a certain part of the EGFR gene
* see if patients whose tumor does shrink with gefitinib treatment are more likely to have a mutation in a certain part of the EGFR gene
* see if the pattern of protein expression in the blood is related to the tumor's sensitivity or resistance to gefitinib treatment.
* see if expression of certain genes in the tumor are related to the tumor's sensitivity or resistance to gefitinib treatment.

DETAILED DESCRIPTION:
This is a phase II, single institution trial to correlate gefitinib response and mutations in the protein-tyrosine kinase domain of the EGF receptor gene. The study will be conducted in patients with Stage I and II NSCLC who have been determined to be operable and resectable.

Patients must have 1 or more of the following features: never smoker or smoking history of < 15 pack years and/or features of bronchioloalveolar lung cancer. 50 patients will be enrolled on this study. Treatment will be with gefitinib for at least 21 days before surgery (depending on the timing of the surgery). Patients will discontinue gefitinib 2 days before their operation. For patients that demonstrate a radiographic response to gefitinib preoperatively and /or patients with mutations in the protein-tyrosine kinase domain of the EGF receptor gene (identified from the surgical sample), gefitinib will continue for 2 years post-surgery. Patients who do not have evidence of radiographic response or mutations in the protein-tyrosine kinase domain of the EGF receptor gene will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of malignancy at Memorial Sloan-Kettering
* Patients must have previously untreated stage I or II NSCLC (T11-2N0M0, T1-2N1M0, T3N0M0) and 1 of the following features: never smoker or < 15 pack year smoking history and/or bronchioloalveolar cancer (either pure BAC, BAC with focal invasion or adenocarcinoma with BAC features)
* Patients must have been determined to be operable and resectable by the treating thoracic surgeon.
* Age >18 years.
* Measurable indicator lesions
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or lactating women or women of childbearing potential not using effective contraception. Men participating in the trial must also use effective contraception when sexually active.
* Patients may not be receiving any other investigational agents.
* Any history of or evidence of interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Dercle L, Fronheiser M, Lu L, Du S, Hayes W, Leung DK, Roy A, Wilkerson J, Guo P, Fojo AT, Schwartz LH, Zhao B. Identification of Non-Small Cell Lung Cancer Sensitive to Systemic Cancer Therapies Using Radiomics. Clin Cancer Res. 2020 May 1;26(9):2151-2162. doi: 10.1158/1078-0432.CCR-19-2942. Epub 2020 Mar 20. PMID 32198149
- [Derived] Zhao B, Oxnard GR, Moskowitz CS, Kris MG, Pao W, Guo P, Rusch VM, Ladanyi M, Rizvi NA, Schwartz LH. A pilot study of volume measurement as a method of tumor response evaluation to aid biomarker development. Clin Cancer Res. 2010 Sep 15;16(18):4647-53. doi: 10.1158/1078-0432.CCR-10-0125. Epub 2010 Jun 9. PMID 20534736
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 65
Completed | 50
Not Completed | 15
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Not completed — Disease Progression | 1
Not completed — Not Treated | 10

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: The Radiographic Response to Gefitinib
Description: Radiographic response is defined as a minor response ( > 25% decrease in the sum of the products of measured lesions)
Time Frame: 21 days
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 50
participants | 21

2. Secondary Outcome: Microarray Analysis to Identify Gene(s) or Gene Clusters That Exhibit Changes in Gene Expression; Time to Relapse and Overall Survival Data
Description: Each patient provides two binary variables: presence/absence of mutation and responder/non responder. The association between the two will be tested using the Fisher's exact test for the resulting 2x2 table.Changes in expression levels within a patient will be assessed using a paired t-test. Similarly differences in expression levels between responders and non-responders will be assessed using a two-sample t-test. Appropriate adjustment will be made for the multiple comparisons problem that arises because there are over 21,000 probe sets on the U133A array.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Groups:
- EGFR Mutation Positive; EGFR Mutation Negative: Tumor specimens analyzed for EGFR mutation
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 17 | 4
percentage of participants
  Disease Free Survival | 85 | 76
  Overall Survival | 98 | 92

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 7/65
Other Adverse Events (participants affected / at risk) | 8/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=65)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Retinopathy (Eye disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=65)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 6 (6)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes